CLINICAL TRIAL: NCT06159608
Title: Sex Differences in the Vascular Effects of E-cigarette Use
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202308025
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: E-cigarette Use
MeSH Terms: conditions — Vaping | interventions — NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Young Women (Other): Young women who do not use e-cigarettes
  Interventions: Drug: Local heating + L-NAME (NG-nitro-L-arginine methyl ester; nitric oxide synthase inhibitor); Other: Chronic estrogen exposure
- Healthy Young Men (Other): Young men who do not use e-cigarettes
  Interventions: Drug: Local heating + L-NAME (NG-nitro-L-arginine methyl ester; nitric oxide synthase inhibitor)
- Young Women using E-cigarettes (Other): Young women chronically use e-cigarettes
  Interventions: Drug: Local heating + L-NAME (NG-nitro-L-arginine methyl ester; nitric oxide synthase inhibitor); Other: Chronic estrogen exposure
- Young Men using E-cigarettes (Other): Young men chronically use e-cigarettes
  Interventions: Drug: Local heating + L-NAME (NG-nitro-L-arginine methyl ester; nitric oxide synthase inhibitor)

INTERVENTIONS:
Drug: Local heating + L-NAME (NG-nitro-L-arginine methyl ester; nitric oxide synthase inhibitor) — Differences in endothelium- and nitric oxide (NO)-dependent dilation between groups
Other: Chronic estrogen exposure — differences in urine estrogen levels across the menstrual cycle between women groups only
  Arms: Healthy Young Women; Young Women using E-cigarettes

SUMMARY:
The use of electronic nicotine delivery systems, or e-cigarettes - colloquially referred to as "vaping" - in the United States has increased exponentially since their introduction to the US market in 2007. Prevalence of ever and current e-cigarette use is highest among teenagers and young adults with 16-28% of this population having reported vaping. While the majority of e-cigarette users are current tobacco smokers, 32.5% of current e-cigarette users are never- or former-smokers, representing a growing population of young adults who exclusively vape. While e-cigarettes have been marketed as a safer alternative to tobacco cigarettes, clinical studies examining these claims are limited. Cardiovascular disease (CVD) is the primary cause of premature death among tobacco cigarette smokers and reductions in vascular endothelial function, a significant predictor of future CVD, are detectible in otherwise healthy young adults who smoke. Despite the explosion in e-cigarette use among young adults, the health effects - especially the effects on mechanisms of vascular function - of these devices remain relatively unexplored.

In this study, we use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) we examine the blood vessels in a dime-sized area of the skin in otherwise healthy young (18-24yrs) chronic e-cigarette users. Local heating of the skin at the microdialysis sites is used to explore differences in mechanisms governing microvascular control. As a compliment to these measurements, we also draw blood from the subjects to measure circulating factors that may contribute to cardiovascular health and examine markers of inflammatory activation. We will also collect urine from female participants to measure estradiol.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old
* one of the following:

  1. have no history of e-cigarette use
  2. be a current e-cigarette user who has been using e-cigarettes for 6 months or longer

Exclusion Criteria:

* history of cardiovascular, metabolic, and/or skin diseases
* body mass index >30 kg/m2
* blood pressure ≥140 systolic and/or ≥ 90 diastolic
* current or history of tobacco cigarette use
* current antihypertensive or cholesterol-lowering medication
* current use of cannabis, marijuana, and/or other illegal substances
* current use of stimulant drugs
* currently pregnant or breastfeeding
* allergy to materials used during the experiment (e.g. latex),
* known allergy to study drugs
* healthy control subjects will also be excluded if they have ever used e-cigarettes in the past

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular endothelium-dependent dilation response measured by laser-Doppler flowmetry | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator responses to local heating over a microdialysis fiber receiving lactated Ringer's solution, followed by L-NAME infusion to quantify NO-dependent response
monthly estrogen exposure | 1 month
  daily estradiol levels will be measured in all women for 1 month/menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No